CLINICAL TRIAL: NCT01261000
Title: Tissue Biomarker for Pegvisomant Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Shlomo Melmed, MD, Executive Vice President, Academic Affairs, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro23051; WS921563 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Results first posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-07

CONDITIONS: Acromegaly
Keywords: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — pegvisomant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pegvisomant (Experimental)
  Interventions: Drug: Pegvisomant

INTERVENTIONS:
Drug: Pegvisomant — Pegvisomant used as indicated
  Other Names: Somavert

SUMMARY:
Acromegaly is a disease of the pituitary gland that involves overproduction of growth hormone. Pegvisomant works by blocking binding of GH to receptors found in tissues throughout the body. Human studies have evaluated pegvisomant action by measuring reduction of IGF-I levels in the blood. However, no studies have evaluated the effects of blocking GH receptors in tissues. In this study, we will study tissue biomarkers for pegvisomant action in GH and IGF-I dependent signaling pathways in colon tissue of patients with acromegaly treated with pegvisomant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acromegaly established on the basis of symptoms and signs at presentation, evidence of a pituitary adenoma on MRI, elevated serum concentrations of IGF1 (>1.3 X ULN), and inadequate GH suppression (>0.4 ng/mL) following OGTT
* Candidates to receive pegvisomant therapy following pituitary adenoma surgery, or intolerant of other medical treatments or had not undergone previous therapy
* Normal LFTs before treatment
* Dynamic testing of the pituitary axis and, if applicable, appropriate hormone replacement

Exclusion Criteria:

* Treatment with a long-acting SRL within 12 weeks before enrollment
* Presence of a macroadenoma with visual field defects as a result of chiasmatic compression
* Clinically significant hepatic abnormalities and/or AST or ALT >3 X ULN on screening
* Known hypersensitivity to any of the test materials or related compounds
* History of, or known current, problems with alcohol or drug abuse
* Any mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study, and/or evidence of an uncooperative attitude

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Melmed, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Chesnokova V, Zonis S, Zhou C, Recouvreux MV, Ben-Shlomo A, Araki T, Barrett R, Workman M, Wawrowsky K, Ljubimov VA, Uhart M, Melmed S. Growth hormone is permissive for neoplastic colon growth. Proc Natl Acad Sci U S A. 2016 Jun 7;113(23):E3250-9. doi: 10.1073/pnas.1600561113. Epub 2016 May 25. PMID 27226307

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pegvisomant
Started | 8
Completed | 7
Not Completed | 1
Not completed — Screen failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pegvisomant
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Effect of Pegvisomant on Colon Tissue p53 Expression
Description: Induction of colon tissue expression of p53, a tumor suppressor, using Western blot analysis, after GH receptor blockade with pegvisomant
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pegvisomant
Number analyzed (Participants) | 7
ng/mL | 330.57 (107.33)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Pegvisomant
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegvisomant (N=8)
Bacterial endocarditis (Cardiac disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size due to rare patient population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes